CLINICAL TRIAL: NCT05558631
Title: Lisa Cohort Study: Longitudinal Study of Health Literacy in the Municipality of Leiria
Brief Title: Longitudinal Study of Health Literacy in the Municipality of Leiria
Acronym: Lisa
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto Politécnico de Leiria (Other)
Responsible Party: Principal Investigator, Sara Dias, Principal investigator, Instituto Politécnico de Leiria
Other Study IDs: Lisa Cohort
Record Dates: First submitted 2022-09-16; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Health Literacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Residents of the municipality of Leiria aged 18 years or more.

SUMMARY:
Health literacy (HL) is a topic of increasing importance todays' ever-changing world. Over the past few decades, HL has gained importance, as it is a factor related to health behaviors and outcomes. In Portugal, the last survey was in 2016 and 61% of the population had a problematic or inadequate level of HL in general. Lisa is a cohort study that will measure HL in the adult population residing in the municipality of Leiria over the next 4 years, with measurements every 2 years. Over the years we will promote activities and interventions adjusted to the needs of Leiria's population. At the end we want to understand the changes during the years and improve the health care provided.

DETAILED DESCRIPTION:
The main aim of this study is to measure HL in the adult population residing in the municipality of Leiria over the next 10 years. As secondary objectives, it is intended to characterize anxiety and depression, metabolic risk, alcoholism, and smoking in the in the same population sample and over the same period. The research design follows a longitudinal, prospective closed cohort study of Leiria's residents during ten years. Strengthening the report of observational studies in epidemiology (STROBE) guidelines were applied in alignment of the research objectives. The frequency of data assessment is set to two years, so participants will be contacted five times during the study. The sample will consist of residents of the municipality of Leiria aged 18 years or over, having been determined a sample size of 4003 (2001 men and 2002 women).

The team that conducted the 1st wave survey will be composed by 32 interviewers, who will be recruited by the Center for Innovative Care and Health Technology (ciTechCare) coordination board through a selection process composed of 2 stages: interview selection plus a theoretical and practical training session. The follow-ups of the cohort were decided to be conducted every two years by call. In the 1st wave a face-to-face interview will be conducted with the Computer Assisted Personal Interview (CAPI) system: all interviewers have a tablet with the software (LimeSurvey) which provided the questionnaire, designed by ciTechCare research team, applied to all subjects. Surveys will be administered online via the LimeSurvey platform at baseline and at 2 years, 4 years, 6 years, and 8 years post baseline (5 waves). The baseline and follow-up surveys will comprise the same battery of validated questionnaires and instruments designed to collect information on sociodemographic, lifestyle aspects (tobacco and physical activity), anthropometric variables, auto-report chronic diseases, metabolic risk, anxiety and depression and HL. It will take approximately 30 minutes to complete the survey.

Metabolic risk is assessed by the Finnish Diabetes Risk Score (FINDRISC), to evaluate symptoms of anxiety and depression we applied the Hospital Anxiety and Depression Scale (HADS) Portuguese validated version and HL will be measured by European Health Literacy Survey Questionnaire (HLS-EU-Q47).

Descriptive statistics (mean, standard deviation, median, minimum, maximum, interquartile range, absolute and relative frequencies) will be computed to describe the cohorts' sociodemographic characteristics. At baseline comparisons between groups (eg with and without anxiety) will be undertaken using t-tests for continuous normally distributed variables or Wilcoxon for continuous non-normally distributed variables. Chi-squared tests will be used for categorical variables, and Fisher's Exact test will be used for categorical variables within smaller sample sizes. Comparison between more than two groups will be performed through one-way analysis of variance (ANOVA) for continuous variables and chi-squared test for categorical variables. Factors significantly associated with any disease group will be included in a logistic regression model for further analysis. The effect of specific conditions on HL will be assessed by linear regression, univariable and then multivariable, controlling for potential confounders and also analyzing potential effect modification. Taking into consideration follow-up, the changes in HL, anxiety and depression will be each evaluated by means of variance analysis with measurement repetition. After checking the statistical model pre-requisites, sociodemographic characteristics will be added by means of linear regression analysis in the final model.

ELIGIBILITY:
Inclusion Criteria:

* The study population will be composed by adults (≥ 18 years old) who are non-institutionalized and living in private households in Leiria.

Exclusion Criteria:

* Residing in hospitals, asylums, military barracks or prisons. Individuals who are unable to speak Portuguese or who reveal an inability to respond to the questionnaire, either directly or through a person who lives with them.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed by adults (≥ 18 years old) who are non-institutionalized and living in private households in Leiria. Because there is no reliable list of households in Portugal, a random selection of points in the map of each location will be performed. Addresses will be selected, and afterwards the "random-walks" will start. Interviewers will register each selected address and, if someone is at home, they will collect information on age and gender of the different people living in that address and will give information about the study. In order to assure the successful data collection, up to three visits to each address (one during the weekend) will be made. At each address, the person whose birthday is closest to the day of the visit (aged 18 years or older) will be selected for the interview and, if available, will be immediately asked to answer the questionnaire.
Sampling Method: Probability Sample
Enrollment: 4003 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2033-01-31 (Estimated); Study Completion 2033-01-31 (Estimated)

PRIMARY OUTCOMES:
Health literacy | Health literacy: measuring change over the next 10 years
  HL will be measured by European Health Literacy Survey Questionnaire (HLS-EU-Q16). HLS-EU-Q16 was developed to measure HL in populations, based on a conceptual framework. Each item in the questionnaire assesses the perceived difficulty of a specific health-related task for the respondent. The HLS-EU-Q16 was translated and validated for Portuguese population. The scale contains 16 items that measure HL. Each item assesses the perceived difficulty of completing a specific health-related task by asking "On a scale from very difficult to very easy, how easy would you say it is to [e.g, find information on symptoms of illnesses that concern you]?" Each item is rated on a 4-point Likert-type scale (1, very difficult; 2, fairly difficult; 3, fairly easy; 4, very easy). A higher difficulty score is assumed with lower HL.

SECONDARY OUTCOMES:
Anxiety and depression | Anxiety and depression: measuring change over the next 10 years
  To evaluate symptoms of anxiety and depression we applied the Hospital Anxiety and Depression Scale (HADS) Portuguese validated version. The HADS is a screening tool to apprehend clinically significant states of anxiety and depression in a non-psychiatric hospital setting. Individual anxiety and depression scores are calculated by summation of the appropriate seven items and thus can range from 0 to 21, with higher scores indicating higher levels of anxiety or depression, respectively. In both subscales, a score between 0 and 7 is "normal," between 8 and 10 "mild," between 11 and 14 "moderate," and between 15 and 21 "severe". Presence of anxiety and depression symptoms is defined when HADS scale is ≥11.
Metabolic risk | Metabolic risk: measuring change over the next 10 years
  Metabolic risk is assessed by the Finnish Diabetes Risk Score-FINDRISC (FINDRISC). FINDRISC is a simple and practical tool originally designed in Finland to identify individuals at high risk of type 2 diabetes mellitus onset, without the need for laboratory tests. The score is based on eight easily identifiable parameters (age, body mass index, waist circumference, hypertension, physical activity level, diet, occurrence of previous hyperglycemia, and family history of diabetes) and provides a measure of the probability of developing diabetes over the next 10 years. Findrisc score varies between 0 and 24. A risk score of 0-14 points indicates a low to moderate risk of diabetes (1-17% chance of diabetes over 10 years). A risk score of 15-20 points indicates a high risk of diabetes (33% chance of diabetes over 10 years). A risk score of >20 points indicates a very high risk of diabetes (50% chance of diabetes over 10 years).

REFERENCES:
- [Derived] Batalha MJ, Gabriel T, Valentim A, Soledade A, Gomes C, Alves B, Dos Santos ES, Passadouro R, Dias SS. Health literacy - study protocol for LiSa cohort study. BMC Public Health. 2024 Jun 29;24(1):1737. doi: 10.1186/s12889-024-19148-8. PMID 38951815